CLINICAL TRIAL: NCT01151163
Title: Evaluation of Sleep Disordered Breathing and Autonomic Dysfunction in Fibromyalgia Through Peripheral Arterial Tonometry
Brief Title: Peripheral Arterial Tonometry (PAT) Evaluation of Sleep in Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Jacob N Ablin, Institute of Rheumatology, Tel Aviv Sourasky medical center
Other Study IDs: 0154-10-TLV
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia, Peripheral arterial tonometry, sleep
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fibromyalgia syndrome (FMS) is characterized by the presence of widespread pain, chronic fatigue and typical sleep disturbances. The purpose of the current study is to investigate the nature of sleep disturbance in FMS, using a novel technology. Peripheral arterial tonometry is a method by which peripheral arterial tone is measured non - invasively using in an ambulatory setup during sleep. The information collected reflects autonomic nervous system function and respiratory changes during sleep. We intend to utilize this technique in order to improve our understanding of the interrupted patterns of sleep in FMS and as a possible biomarker which may be used in the future to follow up FMS patients and their response to treatment.

DETAILED DESCRIPTION:
Fibromyalgia Syndrome (FMS) is a clinical entity characterized by the presence of chronic, widespread pain and tenderness throughout the musculoskeletal system. FMS is considered to be a prototype of central pan syndromes, conditions in which augmentation of pain processing by the central nervous system in a major feature (1;2). As such, FMS overlaps with a number of similar "functional" disorders, including TMJD, IBS, Interstitial cystitis, Gulf war syndrome, chronic fatigue syndrome etc (3-5).

A major clinical feature of FMS is the presence of chronic fatigue, which is typically accompanied by a severely disrupted sleep pattern. Difficulty falling asleep, frequent awakening and non-refreshing sleep are all features classically reported by FMS patients. In addition, a number of classic sleep disturbances have been identified among FMS patients such as alpha - wave intrusion, disrupting normal stage IV sleep, as well as nocturnal falls in oxygen saturation (6). Notably, disturbed sleep may contribute not only to chronic fatigue, but also to enhanced pain processing as well as depression in FMS patients (7). Thus, pain inhibitory functions of the CNS, such as the process of Diffuse Noxious Inhibitory Control (DNIC) appear to be impaired in by sleep disruption (8).

Considerable interest has focused on the role of sleep apnea in FMS, as a possible factor contributing to fatigue and pain. Overt obstructive sleep apnea has been diagnosed in some patients (9) while more subtle disruptions of upper airway dynamics, such as increased upper airway pressure, not leading to total airway collapse, has been detected in many patients (10). Other researchers however have challenged the association of FMS with sleep apnea (11).

Autonomic dysfunction is another important clinical manifestation of FMS with common symptoms including presyncope / syncope, palpitations on standing and dizziness (12). Postural Orthostatic Tachycardia Syndrome (POTS) is another autonomic disorder which clinically overlaps with FMS (13).

Traditional polysomnography is a time-consuming and costly procedure, and hence, relatively few FMS patients are formally evaluated for sleep disorders in clinical practice.

The Watch-PATTM100 is a non-invasive device, which utilizes peripheral arterial tone (PAT), reflecting changes in autonomic nervous system function, as a marker for identifying and documenting respiratory disturbances during sleep. The PAT signal is acquired through a non-invasive probe attached to the finger during the sleep. Parameters measured include oxygen saturation, heart rate, sleep and wake states, REM and non-REM sleep.

The purpose of the current study is to use Peripheral Arterial Tonometry (PAT) in order to compare both disturbed sleep breathing and autonomic dysfunction in fibromyalgia patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Fibromyalgia group:

* Patients over 18 years of age
* Fulfilling ACR 1990 criteria for classification of Fibromyalgia

Exclusion Criteria:

* Patients treated with benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from fibromyalgia recruited from the Tel Aviv Sourasky Medical center fibromyalgia clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob N Ablin, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Tel Aviv Sourasky medical center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv